CLINICAL TRIAL: NCT04871698
Title: Improved AD/ADRD Assessment Sensitivities Using a Novel In-Situ Sensor System
Brief Title: On Site Sensors Monitoring Impacts of Cognitive Decline on ADLs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Texas A&M University (Other); Baylor Research Institute (Other); Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, John Fitch, Principal Investigator, National Institute on Aging (NIA)
Other Study IDs: R44AG065118 (NIH)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Dementia; Dementia Alzheimers
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to compare the effectiveness of a continuous monitoring system to assess Activities of Daily Living (ADLs) over time compared to the traditional assessments used by medical professionals as Alzheimer's Disease and Alzheimer's Disease Related Dementias (AD/ADRD) progresses.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English to understand and sign the consent or assent documents.
* Adult over 65 years of age with no children under 18 years old living in residence.
* Adult anticipates they will be living primarily at designated residence over next 18 months.
* Must receive caregiver interaction at least 6 hours/week.
* Must undergo a Mini-Mental State Exam (MMSE) assessment at baseline during recruitment as well as at the end of the study with a resulting score of 11-25 as part of the recruitment phase of the study.
* Must be willing to have home or facility equipped with sensors to obtain activity and location data.

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults 65 and older with mild to moderate dementia.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Demonstrate equivalency of the proposed IoT system against ADCS-ADL/23 Assessment | 18 months
  The ADCS-ADL/23 assessment will be utilized to measure changes in activities of daily living in the sample population while BC's system is also in place independently measuring the changes in activities of daily living.
Identify improved sensitivities for detection of early and moderate-stage AD/ADRD activities of daily living changes | 18 months
  AI techniques will search sensor data for subfactor and novel groupings for statistically significant improvements from what is measured by the ADCS/ADL-23 assessment of decline.

SECONDARY OUTCOMES:
Establish initial data sets and protocols for use of the developed ADL/IADL system data for integration with AD/ADRD research | 18 months
  Database structures and meta-data will be established for anonymous data sets.

CONTACTS AND LOCATIONS:
Locations (1):
- Birkeland Current, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided